CLINICAL TRIAL: NCT06687837
Title: Phase I Trial of Autologous Induced Pluripotent Stem Cell-derived Dopaminergic Progenitor Cell Transplantation for Parkinson's Disease
Brief Title: Treating Parkinson's Disease Through Transplantation of Autologous Stem Cell-Derived Dopaminergic Neurons
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey S. Schweitzer, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey S. Schweitzer, MD, PhD, George A. Lopez, MD Endowed Chair in Neurosurgery, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001089
Record Dates: First submitted 2024-10-24; First posted 2024-11-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Open label, two dosage tiers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose administration (Experimental): 4 million autologous dopaminergic cells will be implanted into the putamen on each side of the brain
  Interventions: Biological: autologous dopaminergic cell implantation
- High dose administration (Experimental): 8 million autologous dopaminergic cells will be implanted into the putamen on each side of the brain
  Interventions: Biological: autologous dopaminergic cell implantation

INTERVENTIONS:
Biological: autologous dopaminergic cell implantation — Dopaminergic progenitor cells derived from autologous induced pluripotent stem cells will be injected into the brain in two cohorts of Parkinson's patients, one receiving low dose and the other high dose (4 and 8 million cells, respectively)

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of the surgical transplantation of dopaminergic progenitor cells into the brains of participants with Parkinson's disease. The transplanted dopaminergic cells will be derived from the participant's own skin cells.

DETAILED DESCRIPTION:
This Phase I, open-label clinical trial aims to assess the feasibility and safety of autologous midbrain dopaminergic progenitor cell (mDAP) transplantation for the treatment of Parkinson's disease. mDAPs will be produced for each participant from a fibroblast sample and then transplanted bilaterally into the putamen under general anesthesia. The study will assess the safety and tolerability of the cell transplant procedure through clinical assessments and neuroimaging (CT, MRI and 18F-DOPA PET) over a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease consistent with the Movement Disorders Society 2015 Parkinson's diagnostic criteria.
* Age 45 - 80 years
* English proficiency sufficient to understand the consent form and participate in a discussion of risks and benefits
* At least 5 years since Parkinson's disease motor symptom onset
* Modified Hoehn and Yahr stage 3-4 in "off"-medication state
* Motor symptoms responsive to levodopa and/or dopamine agonist, defined as taking at least 300 mg/day of levodopa and exhibiting improvement between "off" and "on" MDS-UPDRS of at least 30%
* At least 3 hours of cumulative "off" time per day
* Stable regimen of Parkinson's medications, including levodopa and dopamine agonists, for at least 4 weeks prior to screening.
* Acceptable surgical laboratory values including:

  1. Platelets > 100×109/L (transfusion independent)
  2. Prothrombin time / partial thromboplastin time in normal range and international normalized ratio ≤ 1.3
  3. Aspartate aminotransferase and alanine aminotransferase < 2.5x the upper limit of normal
  4. Serum creatinine ≤ 1.5mg/dL
  5. White blood cell count < 12×109/L.
  6. Estimated glomerular filtration rate ≥ 30 mL/min/1.73m2
* Subject agrees to defer elective neurological surgery, including deep brain stimulation or lesional procedure for PD, invasive treatments, including levodopa or apomorphine infusion, or pump- pump-administered levodopa intestinal gel, until after the study's primary outcome is completed.
* Findings on baseline 18F-DOPA PET imaging consistent with dopaminergic denervation of the putamen
* Subject is willing and able to comply with all study visits and procedures in the opinion of the Investigator.

Exclusion Criteria:

* Subjects unable to give consent due to dementia or psychosis.
* Montreal Cognitive Assessment (MoCA) score < 26
* Subjects with a first-degree relative with Parkinson's disease or with a known genetic mutation predisposing to the development of Parkinson's disease (i.e. this initial study is confined to the more common "sporadic" vs a "genetic" form of the disease).
* Atypical Parkinsonism (Parkinson's-Plus syndrome, secondary parkinsonism)
* Moderate or severe levodopa-induced dyskinesias in any body segment (such patients were found to be more prone to graft-induced dyskinesias in the fetal tissue studies that are proof of priniciple for this therapy)
* Neurologic history or imaging demonstrating brain pathology not directly related to Parkinson's disease that is likely to interfere with study compliance or assessment of Parkinson's related motor disability.
* History of stroke or transient ischemic attack
* History of subarachnoid hemorrhage
* Presence or history of psychosis within 12 months of screening
* Suicidal ideation associated with intent or plan in the past 12 months (an answer of "yes" to C-SSRS questions 4 or 5) or with a previous history of suicide attempts in the past 5 years.
* History of intracranial surgery including deep brain stimulation, focused ultrasound, stereotactic or radiosurgical lesion therapy
* History of malignancy within 5 years. Exceptions will be made for treated cutaneous squamous cell or basal cell carcinoma without evidence of metastasis.
* Use of anticoagulation / antiplatelet agents that cannot be stopped for one week in advance of and two days following surgery without significant risk to the subject
* Use of chronic immunosuppressive therapy including chronic steroids
* Contraindication to MRI or MRI contrast agents
* Pregnant or nursing women
* Subjects with active cardiovascular and cerebrovascular disease within 6 months prior to signing the informed consent form.
* History of severe heart failure (congestive heart failure of New York Heart Association Class II or above or left ventricular ejection fraction < 35% by any examination method), unstable angina pectoris and myocardial infarction/
* Severe arrhythmia
* History of cardiovascular surgery (cardiac, vascular stent surgery, angioplasty)
* Patients with major vascular diseases (aortic aneurysm, aortic dissecting aneurysm, internal carotid artery stenosis)
* Hypertensive patients with poorly controlled blood pressure (defined as blood pressure consistently above 160/100 mmHg despite treatment with antihypertensive drugs) and patients with severe postural hypotension
* Diabetic patients with poorly controlled blood glucose (glycosylated hemoglobin > 9.0%, or fasting plasma glucose (FPG) ≥ 11.1 mmol/L);
* Subjects with alcohol or drug addiction

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 years from time of implantation
  Incidence and severity of adverse events and serious adverse events

SECONDARY OUTCOMES:
18-F DOPA PET uptake | 2 years from time of implantation
  Change in putaminal 18F DOPA PET uptake from baseline to 12 and 24-month follow-up.
Change in motor function | 2 years from time of implantation
  Change in the on-state and practically defined off-state motor function as assessed by the MDS-UPDRS part III from baseline to 12 and 24-month follow-up.
Change in "off" hours | 2 years from time of implantation
  Change in the number of waking hours spent in the "off" state as measured using a self-reported symptom diary, comparing baseline to 12 and 24-month follow-up.
Change in dyskinesia | 2 years from time of implantation
  Change in the frequency and severity of dyskinesia as assessed by the MDS-UDysRS from baseline to 12 and 24-month follow-up.
Change in PD medication usage | 2 years from time of implantation
  Change in the Parkinson's disease medication usage as defined by the levodopa equivalent daily dose (LEDD) from baseline to 12 and 24-month follow-up.
Change in Parkinson's disease related quality of life | 2 years from time of implantation
  Change in the Parkinson's disease-related quality of life as assessed by the change in PDQ-39 from baseline to 12 and 24-month follow-up.
Global impression of change | 2 years from time of implantation
  Patient and Clinician Global Impression of Change (PGI-I and CGI-I) assessed at 12 and 24-months after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States